CLINICAL TRIAL: NCT04131101
Title: Housing Conditions: Evaluation, Advocacy and Research in Toronto Community Housing
Acronym: HEARTH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SMH-18-154
Record Dates: First submitted 2019-05-31; First posted 2019-10-18 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Housing
Keywords: Community organizing; Advocacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Community Organizing (Experimental): All tenants in three TCHC buildings will be invited to participate in a survey on their building conditions at baseline, 6 months and 12 months. Once baseline data collection is complete, there will be a community organizing campaign involving tenants to advocate for improved building conditions.
  Interventions: Behavioral: Community Organizing

INTERVENTIONS:
Behavioral: Community Organizing — The intervention will be community organizing and will consist of engaging tenants, health providers, legal service staff, social service agencies and advocacy organizations (e.g. ACORN). Each building team will identify initial priorities and then invite all building members to discuss and to finalize, as well as a plan for change. Building teams will engage in advocacy to TCHC and its representatives, and other city departments as appropriate. Engaging in advocacy will consist of a wide range of activities but essentially means presenting evidence (e.g. personal experiences, data) to policymakers and decision makers to affect change.

SUMMARY:
This project will examine whether a health promotion campaign using community organizing and joint advocacy by a coalition of tenants, health providers, social service agencies and advocates can lead to improvements in building conditions and health in social housing.

DETAILED DESCRIPTION:
This community based participatory research project will bring together patients of the St. Michael's Hospital Academic Family Health Team (FHT) who are tenants of Toronto Community Housing Corporation (TCHC) with health providers, legal service staff at the Health Justice Program, social service agencies and advocacy organizations to advocate to improve building conditions in three TCHC buildings. The researchers will evaluate the acceptability and feasibility of this health promotion campaign as well as changes in the state of housing and self rated physical and mental health of tenants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Living in one of the three TCHC buildings

Exclusion Criteria:

* under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
Tenant engagement in intervention | 12 months
  Acceptability and feasibility of the intervention, assessed through qualitative focus groups with participants in each intervention building. The HEARTH Survey was built by the research team (example question: How satisfied are you with the condition of your building?). All qualitative data will be managed and analyzed with the data management software, NVivo.
Building conditions | 12 months
  Change in the state of housing evaluated by a questionnaire completed by tenants and official reports from the Toronto Community Housing Corporation. The HEARTH survey consisted of various questions relating to this, leading to different answers due to different scales. For example, for safety of the building, the options were: very safe, fairly safe, neither safe nor unsafe, fairly unsafe, and very unsafe. All scales had 5 options/outcomes but different wordings. No quantitative score was used for this.
Health (Patient-Reported Outcomes Measurement Information System (PROMIS) scale) | 12 months
  Change in self-rated physical and mental health, sense of security, social integration, evaluated by surveys of residents using PROMIS scale. This scale is validated. For pain, the minimum score is 0 and the maximum score is 10, with 10 representing the worst pain imaginable. The higher the number on the scale, the worse the outcome/issue is.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Pinto, MSc MD, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided